CLINICAL TRIAL: NCT02962375
Title: Pilot Study to Assess the Effect of Orange Pomace Fiber on Glycemic Response in Healthy Adults
Brief Title: Effect of Orange Pomace Fiber on Glycemic Response
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2016-118
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: orange pomace fiber; glycemic response
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): 100% orange juice with orange pomace fiber
  Interventions: Dietary Supplement: Active
- Control Treatment (Placebo Comparator): 100% orange juice
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Active — 100% orange juice with orange pomace fiber
  Arms: Active Treatment
Dietary Supplement: Control — 100% orange juice
  Arms: Control Treatment

SUMMARY:
Primary object is to determine if 100% orange juice with enzyme-treated orange pomace fiber compared to a 100% orange juice will reduce 2 hr glycemic response as measured by glucose area under the curve.

Secondary object is to assess if 100% orange juice with enzyme-treated orange pomace fiber compared to a 100% orange juice will reduce 2 hr insulin iAUC response.

DETAILED DESCRIPTION:
The study is single-center, randomized, 2-arm, and crossover design. Twelve healthy men and women aged 20-45 will be recruited for the study. Interested subjects will be asked to come to the Clinical Nutrition Research Center (CNRC) on the IIT Campus, Chicago, IL, where the study will take place for a screening visit to determine if they are eligible to participate in the study. The screening visit will take 2-2.5 hours. Prospective subjects must read, sign and date a written Institutional Review Board (IRB) approved Informed Consent Form prior to performing any study procedure.

At the on-site screening visit, subject will be asked to arrive after overnight fasting for 10-12 hours and be well-hydrated. Subject will be instructed to aim for a water intake of at least 8-10 cups for the 24 hours before the screening visit. Determine eligibility to participate includes having subjects to complete a series of questionnaires related to their health, medication use, dietary habits, and physical activity history. Anthropocentric (height, weight and waist circumference), ear temperature, and vital signs (blood pressure and heart rate) will be measured. Body mass index (BMI) will be calculated from height and weight measurements. BMI is an estimate of body fat based on height and weight that applies to both adult men and women. Fasting blood glucose level by capillary blood from finger prick will be tested. For vital sign measurements, subjects will sit in a comfortable chair, feet uncrossed and on the floor and will be asked to rest quietly for 5 minutes before measuring blood pressure and heart rate. Arm vein will be assessed using a vein access scale test. Subject will be instructed to complete a 24-hour food recall.

Based on the results of the questionnaires, BMI calculation, health evaluation and 24-hour food recall, subjects who meet the inclusion and exclusion criteria will be invited to participate in the study. Eligible subjects will be trained and instructed to record all food and beverages consumed for a 3-day period on food record diaries. Study staff will provide the food record forms and training to the subjects.

Eligible participants will be asked to come to the center for two test days. Test Day 1 will follow the screening visit by at least a 7 day washout adhering to diet instructions.

At each Test Day visit, subjects will arrive at the clinic between 7 am and 9 am after fasting for 10 to 12 hours and in a well-hydrated and well-rested state. If they are taking medication(s) each morning, they will be asked not to take the medication(s) at home and instead to bring to the clinical nutrition center to be taken in the presence of the study investigator so the medications(s) is taken at the same time before each Study Day visit.

Study protocol adherence will be corroborated by asking about the period of fasted state. Subject will also be asked about their limitation/avoidance of polyphenolic diet the last one week and detailed food intake the 24-hour period prior to the visit to ensure consistency and compliance with the protocol requirements. Subjects experiencing unusual stressful events (such as loss of job, loss of loved one, divorce, etc…) will be rescheduled to a later time agreed upon by the subject and investigator. Subject will be asked about their medication intake and health status since their last visit to ensure that subjects are maintaining their good health and medication intake.

After confirming compliance with protocol, anthropometric measurements and vital signs (blood pressure, heart rate and ear temperature) will be taken. A finger prick for fasting blood glucose will be taken to confirm if subject is fasting. A licensed healthcare professional (LHCP) will evaluate and place a catheter on antecubital site of subject's non-dominant arm. A catheter is a thin flexible tube that allows sampling of blood through one port throughout the Study Day. Once the catheter is placed, a baseline blood sample will be taken (Time point T -5). Subject will be asked to rest for 5 minutes, and then another baseline blood sample will be taken (T 0). After completing 2 baseline blood sampling, subjects will receive a serving of 100% orange juice or 100% orange juice with orange pomace fiber based on computer generated randomization sequence. The randomization sequence will be assigned to each subject on the first Study Day visit (Test Day 1). Additional blood samples will be taken at 15, 30, 45, 60, 75, 90, 105 and 120 minutes after the start of the orange juice. Subjects are allowed to drink water after 60 min and the amount will be recorded. After completion of all study procedures and data/sample collection for the day, the catheter will be removed and subjects will be evaluated for safety and/or discomfort/symptoms before leaving the study site. They will be given a snack and written instructions in preparation for the next visit. Study day visits will be scheduled at least 3 days apart, but not more than 7 days. Test Day 2 will be exactly the same as Test Day 1 except the treatment, which will be the other of 100% orange juice or 100% orange juice with orange pomace fiber based on computer generated randomization sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 20-45 years of age, inclusive.
2. Subject has a BMI of 20.0-24.9 kg/m2, inclusive and weight ≥ 110 lb. at screening visit.
3. Subject is willing to maintain his/her usual physical activity pattern throughout the study period.
4. Subject is willing to follow study instructions including compliance with consumption of study beverage, and study visit schedule.
5. Subject is judged to be in good health on the basis of the medical history.
6. Subject is willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to and during study visits. Vigorous physical activity is defined as an activity requiring a large amount of effort, causing rapid breathing and a substantial increase in heart rate (e.g., running, fast cycling, and fast swimming).
7. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator/s and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has fasting glucose ≥100 mg/dL.
2. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at screening visit.
3. Subject has had major trauma or a surgical event within 2 months of the study.
4. Subject has had a weight change ≥4.5 kg within 2 months of visit.
5. Subject has a history or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary, or gastrointestinal disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
6. Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
7. Subject has a history of extreme dietary habits, as judged by the Investigator (e.g., Atkins diet, etc.).
8. Subject is a vegan or a vegetarian.
9. Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
10. Subject has a known intolerance or sensitivity to any ingredients in the study products.
11. Subject has used medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, hypoglycemic medications, and systemic corticosteroids 2 weeks prior to visit 1 and throughout the study.
12. Subject is a female, who is pregnant, planning to be pregnant during the study period or lactating.
13. Subject is a current smoker. Past smoker abstinence for less than 2 years.
14. Subject has participated in any clinical trial within 30d prior to enrollment.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Changes in plasma glucose concentration as measured by iAUC over a 2 hour Postprandial Test day after administration of active treatment compared to control treatment | 2 hours
  plasma glucose concentration as measured by iAUC over a 2 hour

SECONDARY OUTCOMES:
Changes in plasma insulin concentration as measured by iAUC over a 2 hour Postprandial Test day after administration of active treatment compared to control treatment | 2 hours
  plasma insulin concentration as measured by iAUC over a 2 hour

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided